CLINICAL TRIAL: NCT02649153
Title: Effect of Smoked Plum and Chewing Gum on Postoperative Bowel Function Following Hepatic Resection
Acronym: SP/GC-HCC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Guangxi Medical University (Other)
Responsible Party: Principal Investigator, Jian-Hong Zhong, Director, Guangxi Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SP/GC-HCC
Record Dates: First submitted 2016-01-05; First posted 2016-01-07 (Estimated); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Liver Cancer
MeSH Terms: conditions — Liver Neoplasms | interventions — Chewing Gum

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- smoked plum (Experimental): Patients will receive smoked plum (3 piece each time, three times per day) starting in the first day after resection until flatus.
  Interventions: Drug: smoked plum
- gum chewing (Active Comparator): Patients will receive gum chewing (three times per day) in the first day after resection until flatus.
  Interventions: Drug: gum chewing
- empty control (No Intervention): This group patients will not receive gum chewing or smoked plum.

INTERVENTIONS:
Drug: smoked plum — Patients will receive smoked plum (3 piece each time, three times per day) starting in the first day after resection until flatus
  Arms: smoked plum
Drug: gum chewing — Patients will receive gum chewing (three times per day) in the first day after resection until flatus.
  Arms: gum chewing

SUMMARY:
Every patient undergoing surgery in the abdomen, such as hepatic resection, will experience temporary paralysis of bowel function. This study aims to evaluate whether smoked plum and chewing gum can reduce the bowel paralysis after hepatic resection in patients with hepatocellular carcinoma. One third of the study population will receive smoked plum, one third with chewing gum, and the last will act as empty control.

DETAILED DESCRIPTION:
Hepatectomy is widely used to treat patients with hepatocellular carcinoma (HCC), even those with intermediate and advanced disease. Despite its well-demonstrated clinical safety and efficacy in many patients, it is associated with postoperative morbidity and mortality. One complication after hepatectomy is delayed resumption of gastrointestinal function, known as postoperative ileus. This can decrease patient comfort and increase morbidity and mortality, prolonging hospital stay and raising healthcare costs. While postoperative ileus usually resolves within approximately 3 days, it can last longer in some cases as a condition termed postoperative paralytic ileus. Postoperative use of opioid-based analgesics can increase incidence of postoperative ileus.

No drugs or interventions to prevent or treat postoperative ileus have been approved by the China Drug Administration or the US Food and Drug Administration. Several studies show that chewing gum, a new and simple modality, can accelerate complication-free recovery of gastrointestinal function following gastrointestinal surgery and obstetrical-gynecological surgery. This raises the question whether postoperative smoked plum, or chewing gum can reduce risk of postoperative ileus following hepatectomy. To examine this question, we conducted a randomized controlled trial to compare incidence of postoperative ileus and length of hospital stay in HCC patients who received smoked plum, chewing gum or no intervention following hepatectomy.

ELIGIBILITY:
Inclusion Criteria:

* Underwent open hepatic resection
* Diagnosis of HCC was confirmed by histopathological examination of surgical samples in all patients

Exclusion Criteria:

* Previously underwent exploratory laparotomy
* Laparoscopic surgery
* Known Central Nervous System tumors including metastatic brain disease
* History of organ allograft
* Substance abuse, medical, psychological or social conditions that may interfere with the patient's participation in the study or evaluation of the study results
* Any condition that is unstable or which could jeopardize the safety of the patient and his/her compliance in the study
* Pregnant or breast-feeding patients

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Time to first peristalsis | 3 days

CONTACTS AND LOCATIONS:
Overall Officials: Le-Qun Li, MD, Principal Investigator — Affiliated Tumor of Guangxi University
Locations (1):
- Affiliated Tumor of Guangxi University, Nanning, Guangxi, China

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] You XM, Mo XS, Ma L, Zhong JH, Qin HG, Lu Z, Xiang BD, Wu FX, Zhao XH, Tang J, Pang YH, Chen J, Li LQ. Randomized Clinical Trial Comparing Efficacy of Simo Decoction and Acupuncture or Chewing Gum Alone on Postoperative Ileus in Patients With Hepatocellular Carcinoma After Hepatectomy. Medicine (Baltimore). 2015 Nov;94(45):e1968. doi: 10.1097/MD.0000000000001968. PMID 26559269
- [Result] Jang SY, Ju EY, Kim DE, Kim JH, Kim YH, Son M, Jang M, Jeong JH, Kim KS. First flatus time and xerostomia associated with gum-chewing after liver resection. J Clin Nurs. 2012 Aug;21(15-16):2188-92. doi: 10.1111/j.1365-2702.2012.04132.x. Epub 2012 Jun 2. PMID 22672009